CLINICAL TRIAL: NCT00888108
Title: A Phase 1 Safety and Pharmacokinetic Study of ABT-263 in Combination With Taxotere® (Docetaxel) in the Treatment of Subjects With Solid Tumors
Brief Title: Safety Profile, MTD, and PK Profile Studies of ABT-263 When Administered in Combination With Standard and Weekly Regimens of Docetaxel in Subjects With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-338; 2008-001477-15 (EudraCT Number)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — navitoclax; Docetaxel

ARMS (1):
- docetaxel +ABT-263 (Experimental)
  Interventions: Drug: ABT-263; Drug: Docetaxel

INTERVENTIONS:
Drug: ABT-263 — 150 mg of ABT-263 is taken orally once daily on Days 1-5 or Days 1-3 of each 21 day cycle. 150 mg of ABT-263 on Days 1-3, 8-10 and 15-17 of each 28-day cycle. This is a dose escalation study, therefore the dose of ABT-263 will change throughout the study.
Drug: Docetaxel — 75 mg/m2 will be given by intravenous infusion on day 1 of each 21 -day cycle. 30 mg/m2 will be given by intravenous infusion on day 1, 8, 15 of each 28 -day cycle.
  Other Names: docetaxel, taxotere

SUMMARY:
This is a Phase 1 open-label study evaluating the safety of ABT-263 when combined with a standard and weekly regimen of docetaxel in subjects who have solid tumors with measurable disease.

ELIGIBILITY:
Inclusion Criteria

* Subject must be greater then or equal to 18 years of age.
* Subject must have a histologically and/or cytologically documented cancer for which docetaxel has been determined to be an appropriate therapy, per the Investigator.
* Subject must have evaluable and/or measurable disease by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) as defined by RECIST.
* Subjects with brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 28 days prior to the first dose of study drug.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of less then or equal to 1.
* Subject must have adequate bone marrow, renal and hepatic function per local laboratory reference range as follows:

  * Bone marrow: Absolute Neutrophil Count (ANC) greater then or equal to 1500/microliters; platelets greater then or equal to 150,000/mm^3; hemoglobin greater then or equal to 9.0 g/dL;
  * Renal function: Serum creatinine less then or equal 2.0 mg/dL or calculated creatinine clearance greater than or equal to 50 mL/min;
  * Hepatic function and enzymes: AST and ALT less then or equal to 1.5 x the upper limit of normal (ULN) of institution's normal range, ALP less then or equal to 2.5 x ULN, and bilirubin less then or equal to 1.0 x ULN. Subjects with bone metastasis may have ALP less then or equal to 5.0 x ULN.
  * Coagulation: aPTT and PT not to exceed less than or equal to 1.2 x ULN.
* Female subjects must be surgically sterile, postmenopausal (for at least one year), or have negative results for a pregnancy test performed as follows:
* At Screening via a serum sample obtained within 14 days prior to initial study drug administration, and
* Prior to dosing via a urine sample obtained on Cycle 1 Day 1, if it has been greater then 7 days since obtaining the serum pregnancy test results.
* Female subjects not surgically sterile or postmenopausal (for at least one year) and non-vasectomized male subjects must practice at least one of the following methods of birth control:

  * total abstinence from sexual intercourse (minimum one complete menstrual cycle);
  * vasectomized partner;
  * hormonal contraceptives (oral, parenteral or transdermal) for at least three months prior to study drug administration;
  * Double-barrier method (including condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream).
* The subject, or legal representative, must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria

* The subject has an underlying, predisposing condition of bleeding or currently exhibits signs of bleeding. The subject has a recent history of thrombocytopenia associated with bleeding within 1 year prior to first dose of study drug.
* The subject is currently receiving or requires anticoagulation therapy or any drugs or herbal supplements that affect platelet function, with the exception of low-dose anticoagulation medications (i.e., Heparin) that are used to maintain the patency of a central intravenous catheter.
* A female subject is pregnant or breast-feeding.
* The subject has active peptic ulcer disease or other potentially hemorrhagic esophagitis/gastritis.
* The subject has active immune thrombocytopenic purpura (ITP), autoimmune hemolytic anemia (AIHA), or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug).
* The subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal therapy (with the exception of hormones for hypothyroidism, estrogen replacement therapy [ERT], anti estrogen analogs, agonists required to suppress serum testosterone levels [e.g., LHRH, GnRH, etc.] for subjects with prostate cancer if on a stable dose for at least 21 days prior to the first dose of study drug), or any investigational therapy with 14 days prior to the first dose of study drug, or has not recovered to less than a grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy.
* The subject has received an antibody therapy or other biologic (with the exception of colony stimulating factors [G-CSF, GM-CSF] or erythropoietin) within 28 days prior to the first dose of study drug.
* The subject has consumed grapefruit or grapefruit products within 3 days prior to the first dose of study drug.
* The subject has received steroid therapy for anti-neoplastic intent within 7 days prior to the first dose of study drug with the exception of inhaled steroids for asthma, topical steroids, replacement/stress corticosteroids, or corticosteroids taken as premedication for this study.
* The subject has received aspirin or known CYP3A inhibitor (e.g., ketoconazole) within 7 days prior to the first dose of study drug.
* The subject has undergone an allogeneic stem cell transplant.
* The subject has received radio-immunotherapy within 6 months prior to the first dose of study drug.
* The subject has a history of hypersensitivity to docetaxel or other polysorbate 80 drugs.
* The subject has tested positive for human immunodeficiency virus, HIV (due to potential drug-drug interactions between anti-retroviral medications and navitoclax (ABT-263), as well as anticipated navitoclax (ABT-263) mechanism based lymphopenia that may potentially increase the risk of opportunistic infections and potential drug-drug interactions with certain anti infective agents).
* The subject has a significant history of cardiovascular (e.g., MI, thrombotic or thromboembolic event in the last 6 months), renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease that in the opinion of the investigator would adversely affect his/her participating in this study. Questions regarding inclusion of individual subjects should be directed to the Abbott Medical Monitor or designee.
* The subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * active systemic fungal infection;
  * A diagnosis of fever and neutropenia within 1 week prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile of navitoclax (ABT-263) when administered in combination with a standard and weekly regimen of docetaxel. | Weekly
Study the pharmacokinetic interaction of navitoclax (ABT-263) and docetaxel | Weekly
Determine the maximum tolerated dose (MTD) of navitoclax (ABT-263) with a standard regimen of docetaxel | Weekly
Determine the MTD of both navitoclax and docetaxel with a weekly schedule. | Weekly

SECONDARY OUTCOMES:
Evaluate safety at the defined recommended Phase 2 dose (RPTD) and schedule in combination with a standard and weekly regimen of docetaxel. | Bimonthly
Evaluate preliminary data regarding progression free survival | Bimonthly
Evaluate preliminary data regarding objective response rate | Bimonthly
Evaluate preliminary data regarding overall survival | Bimonthly
Evaluate preliminary data regarding duration of overall response | Bimonthly
Evaluate preliminary data with Eastern Cooperative Oncology Group (ECOG) performance status | Bimonthly
Evaluate biomarkers | Bimonthly
  Define the relationship between disease states, B-Cell Lymphoma 2 (Bcl-2) family protein expression, and potential response to the proposed therapy navitoclax when added to a standard and weekly regimen of docetaxel.

CONTACTS AND LOCATIONS:
Overall Officials: Mack Mabry, MD, Study Director — Abbott
Locations (6):
- United States (3):
  - Site Reference ID/Investigator# 51982, Scottsdale, Arizona
  - Site Reference ID/Investigator# 44182, Fort Lauderdale, Florida
  - Site Reference ID/Investigator# 43962, Baltimore, Maryland
- Netherlands (2):
  - Site Reference ID/Investigator# 12844, Rotterdam
  - Site Reference ID/Investigator# 20042, Rotterdam
- Site Reference ID/Investigator# 12845, Surrey, United Kingdom

REFERENCES:
- [Derived] Puglisi M, Molife LR, de Jonge MJ, Khan KH, Doorn LV, Forster MD, Blanco M, Gutierrez M, Franklin C, Busman T, Yang J, Eskens FA. A Phase I study of the safety, pharmacokinetics and efficacy of navitoclax plus docetaxel in patients with advanced solid tumors. Future Oncol. 2021 Jul;17(21):2747-2758. doi: 10.2217/fon-2021-0140. Epub 2021 Apr 14. PMID 33849298